CLINICAL TRIAL: NCT05798910
Title: Comparing the Outcomes of Virtual Reality Based Serious Gaming and Lecture Based Training for Advanced Life Support Trainings: Randomized Control Trial
Brief Title: Comparing the Outcomes of Virtual Reality Based Serious Gaming and Lecture Based Training for Advanced Life Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Emin Aksoy, Principal Investigator, Assoc.Prof.Dr., Director of Medical Simulation Center, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-19/04
Record Dates: First submitted 2023-03-10; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Advanced Cardiac Life Support
Keywords: Advanced Cardiac Life Support; Virtual Reality; Serious Game

STUDY DESIGN:
Intervention Model Description: The members of the conventional group had to complete pretest at the beginning of the study. Afterwards they had to take part at an interactive classroom based lecture about ALS. The next step was the skills training with task trainers in order to teach them compression skills. Afterwards, the conventional group was divided into three blue code teams consisting of each 5 participants for the simulation session. Two independent instructors evaluated the video recordings in terms of technical and nontechnical skills. The final stage of the study were completing the post-test. The members of VR group had a similar study flow but they had to play with the VR based ALS serious game module instead of the theoretical lecture. A survey about preference of VR based trainings was conducted for the members of the VR group. Mann Whitney U Test and Wilcoxon Signed Ranks Test were used for statistical analysis of the two groups' performances in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Training Group (15 Participants) (Active Comparator): The members of the conventional group had to complete pretest at the beginning of the study. Afterwards they had to take part at an interactive classroom based lecture about Advanced Life Support. The next step was the skills training with task trainers in order to teach them compression skills. Afterwards, the conventional group was divided into three blue code teams consisting of each 5 participants for the simulation session. Two independent instructors evaluated the video recordings in terms of technical and nontechnical skills. The final stage of the study were completing the post-test.
  Interventions: Other: Lecture based training for advanced life support
- VR Group (14 Participants) (Active Comparator): The members of the VR group had to complete pretest at the beginning of the study. Afterwards they had to play with the VR based serious game module for Advanced Life Support. The next step was the skills training with task trainers in order to teach them compression skills. Afterwards, the conventional group was divided into three blue code teams consisting of each 5 participants for the simulation session. Two independent instructors evaluated the video recordings in terms of technical and nontechnical skills. The final stage of the study were completing the post-test. The aprticipants of this group were also asked to fill a survey about their VR experience during the study.
  Interventions: Other: ALS VR (VR based serious gaming module for advanced life support training)

INTERVENTIONS:
Other: ALS VR (VR based serious gaming module for advanced life support training) — Using VR based serious gaming module for advanced life support training instead of taking part in a classical lecture about advanced life support.
  Arms: VR Group (14 Participants)
Other: Lecture based training for advanced life support — Taking part in a classical lecture about advanced life support.
  Arms: Conventional Training Group (15 Participants)

SUMMARY:
The hypothesis of this study is to reveal whether virtual reality(VR) based Advanced Life Support(ALS) serious game module can replace classroom-based ALS lecture, which is part of existing ALS training protocol in addition to skills training.

DETAILED DESCRIPTION:
The participants consisting of students from Acibadem Mehmet Ali Aydinlar University Vocational School for Anesthesiology (N=29) were randomly divided into two groups with 15 (Conventional training group) and 14 (VR based training group) participants each. The members of the conventional group had to complete pretest at the beginning of the study. Afterwards they had to take part at an interactive classroom based lecture about ALS. The next step was the skills training with task trainers in order to teach them compression skills. Afterwards, the conventional group was divided into three blue code teams consisting of each 5 participants for the simulation session. Two independent instructors evaluated the video recordings in terms of technical and nontechnical skills. The final stage of the study were completing the post-test. The members of VR group had a similar study flow but they had to play with the VR based ALS serious game module instead of the theoretical lecture during the study flow. A survey about preference of VR based trainings was conducted for the members of the VR group. Mann Whitney U Test and Wilcoxon Signed Ranks Test were used for statistical analysis of the two groups' performances in this study.

ELIGIBILITY:
Inclusion Criteria:

* Having normal or corrected to normal vision
* No history of visually induced motion sickness

Exclusion Criteria:

* Previously experienced VR-induced motion sickness
* Other medical conditions (Epilepsy, vertigo attacks)

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Providing theoretical knowledge about Advanced Life Support Protocol by using VR based serious game module and classroom based theoretical lecture. | 4 hours
  In the beginning of the study, the participants of the two groups (VR Group and Conventional Training Group) have answered the questions of the pretest. Afterwards, one group had VR based training and the other group had classroom based training. After completing the posttest at the end of the study, the pretest and posttest results were evaluated in order to compare the effectivity of VR based training and classroom based training. The maximum score that could be earned from the pretest and posttest 100.
Potential of VR based training to replace classroom based lectures for advanced life support trainings. | 4 hours
  Depending on the comparison of the pretest and posttest results, the participants, who were trained with VR based serious gaming module has similar results compared with the participants, who were trained with a classroom based lecture. The potential of VR based ALS trainings to replace classroom based lecture to provide ALS knowledge was investigated.

OTHER OUTCOMES:
VR preference | 30 minutes
  At the end of the study, the participants of the VR group were asked to fill a survey about their VR experience during the study. The survey for the VR group also revealed that the majority participants would prefer VR based ALS serious gaming module instead of lecture-based educations in the classroom. A five point Likert scale was used in the survey to evaluate the answers of the participants..

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University CASE (Center of Advanced Simulation and Education), Istanbul, Non-US/Canada, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aksoy ME, Ozkan AE, Kitapcioglu D, Usseli T. Comparing the Outcomes of Virtual Reality-Based Serious Gaming and Lecture-Based Training for Advanced Life Support Training: Randomized Controlled Trial. JMIR Serious Games. 2023 Sep 28;11:e46964. doi: 10.2196/46964. PMID 37768719